CLINICAL TRIAL: NCT02036190
Title: Ancillary T Cell Based Studies in SPIROMICS
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: R01HL110883-01A1 (NIH)
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Smoke Induced Lung Disease
Keywords: COPD, chronic obstructive pulmonary disease, emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Former or current smokers without emphysema
- Emphysema: Current or former smokers with emphysema

SUMMARY:
The long-term objectives of this ancillary application are to characterize a subpopulation of smokers with auto-reactive T cell response, to validate immunodiagnostic assays that could detect emphysema, and to find molecular signatures for pathogenic T cell development in a well-characterized cohort participating in SPIROMICS (UCSF center).

DETAILED DESCRIPTION:
One of the major medical challenges facing us is that susceptibility to smoking-induced lung diseases varies greatly and essentially precludes our ability to predict which smokers will develop emphysema. Because the SPIROMICS study is designed to phenotype a large and heterogeneous group of smokers, we have chosen this cohort to identify the subpopulation who have auto-reactive T cells, as this may represent a contributing mechanism in the development of emphysema, which may need alternative therapies, and may represent a group of patients who will have progressive disease despite smoking cessation. In Aim 1, we will prospectively determine the presence of auto-reactive T cell responses as determined by increased cytokine release in 180 ever-smokers with and without emphysema; in Aim 2 we will focus on the longitudinal aspect of the factors that could predispose development of auto-reactive T cells in the population at risk. These studies form the prerequisite basis for developing additional novel immune-based diagnostic and therapeutic strategies in human emphysema. The short-term objectives outlined here are based on our preliminary data, and provide the necessary platform that will be used to answer the following urgent questions: i) in a distinct prospective cohort of ever smokers, can auto-reactive T cells predict the presence of radiographic emphysema? ii) Can we identify unique and persistent transcriptional signature(s) that are associated with autoimmune emphysema? The observational and longitudinal design of SPIROMICS allows for detailed assessment of the association between emphysema as the primary clinical endpoints and could validate the novel T cell specific immunodiagnostic potential that has been developed in our laboratory. We propose to explore the role of autoimmunity as a contributing mechanism in the development of emphysema with the additional aim of bringing current technologies to bear on clinical and future diagnostic tests. PUBLIC HEALTH RELEVANCE: We have discovered specific autoreactive T cells in ever-smokers with emphysema and there is growing evidence linking these particular effector cells with the pathophysiology of smoking related lung disease. Our proposed studies are important because they will provide new diagnostic and prognostic assays (e.g. gamma-6-Spot, based on Th1 and Th17 cytokines) in ever-smokers who have, or are at risk of developing emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Over 4o, former or active smokers

Exclusion Criteria:

* HIV infection, chronic hepatitis B and C, immune suppressive medications.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former or current smokers, over 40 years of age recruited in SPIROMICS at UCSF
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Autoreactive T cell response to elastin fragments | One year
  We will examine cytokines released by T cells in response to elastin fragments

CONTACTS AND LOCATIONS:
Overall Officials: Laura Koth, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No